CLINICAL TRIAL: NCT04121390
Title: Accessing the Effectiveness of a Pediatrician-led Newborn Parenting Class on Maternal Newborn Care Knowledge, Anxiety and Confidence
Brief Title: Assessing the Impact of Mount Sinai Parenting Center's Newborn Class
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Dani Dumitriu, Assistant Professor of Pediatrics and Psychiatry, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 18-0778
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Parenting Intervention
Keywords: Newborn care; Maternal anxiety; Maternal self-efficacy; Newborn care knowledge; Developmental trajectory; Positive parenting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newborn Parenting Class: New Mother who attended the Newborn Parenting Class
  Interventions: Behavioral: Newborn Parenting Class
- New Mothers: New Mothers who expressed interest, but did not attend the Newborn Parenting Class

INTERVENTIONS:
Behavioral: Newborn Parenting Class — Newborn Parenting Class designed by Mount Sinai Parenting Center. The class is 1-hour long and taught be pediatric attending and residents to all families who deliver well babies at Mount Sinai.
  Groups: Newborn Parenting Class

SUMMARY:
This study is the first to evaluate the effectiveness of a Newborn Parenting Class designed by Mount Sinai Parenting Center. The study measures how effective the class is in improving maternal knowledge on newborn care, decreasing maternal self-perceived anxiety and increasing maternal confidence.

DETAILED DESCRIPTION:
The important role positive parenting plays in promoting a child's developmental trajectory has led to the design and implementation of many postpartum education initiatives. With 99% of babies in the U.S. born in hospitals, there is a uniqueness of being in the hospital for an extended period of time with the opportunity to educate parents on the importance of promoting early development. Pediatricians are uniquely well-positioned to address both medical and developmental concerns parents may have during critical periods in a child's development, yet very few interventions are led by pediatricians. The Mount Sinai Parenting Center designed the Newborn Parent Education and Discharge Class (hereafter referred to as Newborn Class) to address this issue. The class is 1-hour long and taught be pediatric attending and residents to all families who deliver well babies at Mount Sinai. The class aims to educate parents about medical issues, responsive parenting, and sleep. It is currently taught every Tuesdays and Thursdays. Because of the limited availability of the class, not all mothers have the opportunity to attend. This research study will survey first time mothers of newborns to explore the effectiveness of attending the class. The study team hypothesizes that attending the class would result in increased knowledge on newborn care, increased confidence levels and decreased levels of anxiety.

First time mothers who delivered a full-term singleton vaginally with no major complications were included in the study. Only mothers who attended the class (intervention) or expressed desire to attend class but were discharged before a class was offered (control) were included in analysis. Mothers were recruited between May 2018 and August 2019 at the Klingenstein Pavilion of Mount Sinai. Maternal self-perceived anxiety and confidence were measured using standardized scales, and knowledge on newborn care was assessed using an internally-developed scale.

ELIGIBILITY:
Inclusion Criteria:

* First-time mother
* Above 18 years old
* Vaginal delivery of a healthy full-term singleton
* No major perinatal complications (per self-report)
* Consent to participate.

Exclusion Criteria:

-none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the study are mothers who delivered vaginally a singleton with no major perinatal complications at Mount Sinai Hospital. Participants were not randomized into control and intervention. This was an Observational study of eligible mothers than attended the Newborn Class ("intervention group") and eligible mothers who wanted to but were not able to attend the Newborn Class because it was not available during their stay at the hospital ("control group").
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory for Adults (STAI) | Immediately after enrollment (Day 1)
  Maternal self-perceived anxiety was measured using State-Trait Anxiety Inventory for Adults (State only). A 40 self-report items questionnaire, each item scored on 4-point likert-type response scale from 1 (not at all) to 4 (almost always), full range from 20 to 80, with higher score STAI scores suggesting higher levels of anxiety
Karitane Parenting Confidence Scale (KPCS) | Immediately after enrollment (Day 1)
  Confidence level was measured using Karitane Parenting Confidence Scale. A 15 item instrument with ach item on the KPCS is scored 0, 1, 2, or 3. Total score range from 0-45, with higher score indicating the parent feeling more confident.
Newborn Care Knowledge Questionnaire | Immediately after enrollment (Day 1)
  Knowledge on newborn care was assessed using an internally-developed scale, developed by a team of pediatricians and specialists.
  Total score ranges from 0-10, with higher score indicating higher level of knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Dani Dumitriu, MD, PhD, Principal Investigator — Columbia University Irving Medical Center; Icahn School of Medicine at Mount Sinai; Blair S Hammond, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).